CLINICAL TRIAL: NCT00486772
Title: Sevelamer, Fetuin-A and Endothelial Dysfunction in CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1-Yilmaz
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-06

CONDITIONS: Vascular Diseases
Keywords: This study was designed to investigate whether the suggested beneficial effects of sevelamer on VC were related to fetuin-A levels in patients with CKD.
MeSH Terms: conditions — Vascular Diseases | interventions — Sevelamer; calcium acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sevelamer (Renagel), calcium acetate (Phos-ex)

SUMMARY:
Vascular calcification and endothelial dysfunction (ED) contribute to the development of cardiovascular disease (CVD) in patients with chronic kidney disease (CKD). Sevelamer, a non-calcium based phosphate binder, has been shown to attenuate cardiovascular calcification in CKD patients while the exact mechanism has not been clarified.

This study was designed to investigate the effect of short-term sevelamer treatment on both serum fetuin-A concentrations and ED seen in CKD patients.

DETAILED DESCRIPTION:
CKD stage 4 patients older than 18 years of age and willing to participate to the study were screened. Those who had serum phosphorus > 5.5 mg/dl were evaluated for the study. Patients with diabetes mellitus, history of coronary artery disease, smokers and those taking statins or renin-angiotensin blockers were excluded because of the effect of these factors on endothelial dysfunction. Of 62 screened patients 50 met the study criteria and were included in this study. Thirty-two healthy subjects were studied as controls. The ethical committee of Gulhane School of Medicine approved the study and written informed consent was obtained from all patients.

Study design:

This was a randomized study conducted from 2005 through 2006 in Gulhane School of Medicine. The Outpatient Clinic of Department of Nephrology is a tertiary referral center. At admission, most patients were untreated (including phosphate binders) or treated only with antihypertensive agents. After the first evaluation, patients receiving phosphate binders (n=9) underwent a 2-week washout period. Patients who developed a phosphate level >5.5 mg/dl during this period were included in the study. Patients were randomly assigned in 1:1 ratio to receive sevelamer (Renagel capsule) or calcium acetate (Phos Ex tablet). The treatment phase was 8 weeks. During the study period serum calcium and phosphorus concentration were measured every 2 weeks and the dose of phosphate binders were titrated to achieve a serum phosphorus concentration < 5.5 mg/dl. The starting dose for sevelamer was 1-2 capsules (800 mg) three times a day and for calcium acetate (1000 mg) 1 tablet three times a day. The medications were given with meal and the doses were increased as needed. Patients were not given calcitriol during the study period.

Fasting blood samples were taken before and after the study to measure serum creatinine, serum albumin, hs-CRP, insulin, iPTH, lipid profile and serum fetuin-A concentration. Additionally, flow-mediated dilatation (FMD) was also evaluated before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 4 patients
* Older than 18 years of age
* Non-diabetic
* Serum phosphorus > 5.5 mg/dl

Exclusion Criteria:

* Diabetes mellitus
* History of coronary artery disease
* Smokers
* Taking statins or renin-angiotensin blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut I Yilmaz, Principal Investigator — Gulhane School of Medicine

REFERENCES:
- [Derived] Caglar K, Yilmaz MI, Saglam M, Cakir E, Acikel C, Eyileten T, Yenicesu M, Oguz Y, Vural A, Carrero JJ, Axelsson J, Lindholm B, Stenvinkel P. Short-term treatment with sevelamer increases serum fetuin-a concentration and improves endothelial dysfunction in chronic kidney disease stage 4 patients. Clin J Am Soc Nephrol. 2008 Jan;3(1):61-8. doi: 10.2215/CJN.02810707. Epub 2007 Dec 5. PMID 18057307